CLINICAL TRIAL: NCT01961440
Title: Prognosis Scoring System for Acute-on-Chronic Liver Failure
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Zhe-bin Wu, Principal Investigator, Third Affiliated Hospital, Sun Yat-Sen University
Other Study IDs: zssywzb02
Record Dates: First submitted 2013-10-09; First posted 2013-10-11 (Estimated); Last update posted 2013-10-11 (Estimated); Status verified 2013-09

CONDITIONS: Liver Failure
MeSH Terms: conditions — Liver Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
This research is to establish a simple and practical system to predict the prognosis of sever hepatitis B.Seven factors (level of serum total bilirubin, prothrombin time, severity of hepatic encephalopathy, hepatorenal syndrome,ascites ,infection and size of liver) which were easier to evaluate and more influential， were included to establish a prognosis scoring system．The scorings of a new score system and MELD were graded at the same time in the patients with sever hepatitis B. And then the distribution figures of survival rates and mortality rates were done according to the scores from low to high. The features of distribution figures of two score system in survival rates and mortality rates and significances of clinical application in certain score were interpreted.

ELIGIBILITY:
Inclusion Criteria:

* serum hepatitis B surface antigen(HBsAg) positive for at least 6 months;
* All patients had a poor general condition, manifested as general malaise, fatigue, jaundice and so on;
* serum T-Bil of 171 mmol/L or more; or serum T-Bil rises 17.1 mmol/L or more per day;

Exclusion Criteria:

* superinfection or co-infection with hepatitis A, C, D, E, cytomegalovirus and HIV, or Epstein-Barr virus;
* other liver diseases such as alcoholic liver disease, drug-induced hepatitis, Wilson disease and autoimmune hepatitis;
* ascites or gastrointestinal bleeding or peptic ulcer or esophageal varix by electronic gastroscope examination;
* decompensated liver cirrhosis;
* severe bacterial or fungal infections;
* a history of diabetes or cardiac disease or hypertension or nephrosis.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The population from large hospitals will be selected.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2013-10; Primary Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
survival rate | twelve weeks